CLINICAL TRIAL: NCT06971042
Title: Early Diagnosis of Acute Respiratory Distress Syndrome (ARDS) in Mechanically Ventilated Patient Using Lung Ultrasound Score in Comparison With CT Chest
Brief Title: Early Diagnosis of ARDS in Mechanically Ventilated Patient Using LUS Score in Comparison With CT
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Roaa Mohamed Ibrahim Elshamy, Resident, Tanta University
Other Study IDs: 36264MS675/8/24
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Acute Respiratory Distress Syndrome; Mechanical Ventilation Complication; Computed Tomography
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Lung Ultrasound — Patients were examined in supine position, using a portable ultrasound machine equipped with a curvilinear transducer (5-3 MHz)
  Other Names: Lung computed tomography

SUMMARY:
The aim of this study is to assess accuracy of Lung ultrasound score for early diagnosis of acute respiratory distress syndrome in patients who expected to be mechanically ventilated more than 24 hour in comparison with computed tomography chest .

DETAILED DESCRIPTION:
Acute respiratory distress syndrome is an acute, diffuse, inflammatory form of lung injury and life-threatening condition in seriously ill patients, characterized by poor oxygenation, pulmonary infiltrates, and acute onset. on a microscopic level, the disorder is associated with capillary endothelial injury and diffuse alveolar damage Acute respiratory distress syndrome is an acute disorder that starts within seven days of the inciting event and is characterized by bilateral lung infiltrates and severe progressive hypoxemia in the absence of any evidence of cardiogenic pulmonary edema. According to the Berlin definition, Acute respiratory distress syndrome is defined by acute onset, bilateral lung infiltrates on chest radiography or computed tomography scan of a non-cardiac origin, and a PaO2/FiO2 ratio of less than 300 mm Hg. The Berlin definition differs from the previous American-European Consensus definition by excluding the term acute lung injury; it also removed the requirement for wedge pressure < 18 mm Hg and included the requirement of positive end-expiratory pressure or continuous positive airway pressure of greater than or equal to 5 cm H20.

Once Acute respiratory distress syndrome develops, patients usually have varying degrees of pulmonary artery vasoconstriction and may subsequently develop pulmonary hypertension. Acute respiratory distress syndrome carries a high mortality, and few effective therapeutic modalities exist to combat this condition Although the Berlin definition of Acute respiratory distress syndrome was a major step forward, some of its limitations were recognized soon after publication. Specifically, it was recognized that its requirement for noninvasive ventilation or invasive ventilation could not be met in settings in which these modalities are not available So consensus conference of 32 critical care develop new global Acute respiratory distress syndrome definition that use high flow nasal oxygen , pulse oximetry in place of arterial blood gas and use of Lung ultrasound to suit limited resource setting .

Lung computed tomography scan is the gold standard in diagnosis of Acute respiratory distress syndrome can provide useful diagnostic information and assess the benefit of treatment. However, this procedure is done in a computed tomography unit under cardiorespiratory monitoring with an increased risk to the patient.

Diagnostic and lung exploratory ultrasound is a rapidly evolving technique used in the Intensive care unit environment, being considered noninvasive, radiation-free, cheap, and easy to perform .

Lung ultrasound has been validated for hemodynamic management, pleural effusions, pulmonary edema, pneumothorax detection, parenchymal consolidation, and central vein catheter placement .

simple and short Lung ultrasound examination could predict prone position oxygenation response in Acute respiratory distress syndrome patients .

Scores based on detection of B-lines (the sonographic sign of increased lung density associated with interstitial syndrome) and on consolidation have been correlated with global and regional lung aeration as assessed by computed tomography chest.

Lung ultrasound has been proposed as an accurate bedside and radiation free technique for evaluation of lung consolidations and for follow-up of aeration changes in response to interventions.

However lung us scoring system hasn't been included in Acute respiratory distress syndrome definition and didn't prefer image modality in diagnosis of Acute respiratory distress syndrome , therefore our study will explore the feasibility and accuracy of lung us score performed bedside to differentiate between Acute respiratory distress syndrome and non Acute respiratory distress syndrome patient compared to lung computed tomography .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 21 years old of both sexes .
* Patients who are expected to be mechanically ventilated more than 24 h .
* Patients who are suspected to be Acute Respiratory Distress Syndrome according to Berlin definition which consists of clinical criteria and with precipitating factors which starts within 1 week of known insult as in trauma patients with lung contusions.

Exclusion Criteria:

* Patient's first guardian who refuse the inclusion in the study .
* History of pre-existing lung disease ( tumors, interstitial lung diseases)
* In cases of volume overload.
* Patients with acute kidney injuiry or renal failure

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted in surgical Intensive care unit that mechanically ventilated more than 24 hours who fulfill criteria of Acute Respiratory Distress Syndrome according to Berlin definition.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of Acute respiratory distress syndrome | Within 48 hours
  Accuracy of lung ultrasound score in diagnosis of Acute respiratory distress syndrome in comparison with Lung computed tomography .

SECONDARY OUTCOMES:
Severity of Acute respiratory distress syndrome . | Within 48 hours
  Accuracy of lung ultrasound score in assessment severity of Acute respiratory distress syndrome .

CONTACTS AND LOCATIONS:
Overall Officials: Roaa Elshamy, MSc, Principal Investigator — Tanta University; Roaa Elshamy, Principal Investigator — Tanta University
Locations (1):
- Tanta university, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
The data will be available upon the reasonable request from the principle